CLINICAL TRIAL: NCT00770289
Title: Open Label, Observational, Non-interventional Study for the Evaluation of Remission Rates in Patients With MDD Under Treatment With Various Anti-depressives
Brief Title: Study Comparing Remission Rates, in Patients With Major Depressive Disorder (MDD)
Acronym: B2411003
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0600B-102374; B2411003 (Other: Pfizer)
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group
  Interventions: Other: Cohort

INTERVENTIONS:
Other: Cohort — Cohort (Patients diagnosed with MDD who are either changing treatment or have never received treatment).

SUMMARY:
Tools known as 'depression scales 'are widely used as assessments to evaluate a patient's response to treatment. The purpose of this study is the evaluation of the remission rates for patients with MDD. The evaluation will involve the use of HAM-D 17, and HAM-D 7 questionnaires and the comparison of those questionnaires.

DETAILED DESCRIPTION:
12 weeks random

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* 18-75 years old
* Patients diagnosed with MDD according to DSM IV without psychotic symptoms
* HAM-D17 > or = 18 on inclusion
* Patients receiving treatment for the first time or changing treatment based on their doctor's decision

Exclusion Criteria:

* Subjects with potentially problematic compliance
* Subjects participating in an interventional trial within the last 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with MDD who are either changing treatment or have never received treatment.
Sampling Method: Probability Sample
Enrollment: 851 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Greece (2):
  - Pfizer Investigational Site, Haidari, Athens
  - Pfizer Investigational Site, Ilissia, Athens

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0600B-102374&StudyName=Study%20comparing%20remission%20rates%2C%20in%20patients%20with%20%20Major%20Depressive%20Disorder%20%28MDD%29

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants diagnosed with major depressive disorder (MDD) who either started treatment with any anti-depressive agent for MDD for the first time or had a change in treatment as per physician's discretion.
Period: Overall Study
Arm/Group | All Participants
Started | 851
Completed | 845
Not Completed | 6
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 851
Age Continuous [Mean (Standard Deviation); unit: years] — Out of 851 participants, data for the baseline measure, age, was available only for 849 participants.
  years | 46.2 (13.2)
Sex/Gender, Customized [Number; unit: participants]
  Female | 528
  Male | 322
  Not available | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Remission Based on Hamilton Depression Scale (HAM-D)
Description: Remission according to HAM-D: HAM-D17 score less than or equal to (=<) 7 or a HAM-D7 score =< 3. HAM-D17: standardized, clinician-administered rating scale; assesses 17 items characteristically associated with major depression. Individual items are scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), with 0=none/absent and 4=most severe. Total score: 0 to 66; higher score indicates more depression. HAM-D7: subset of HAM-D17; assesses 7 items associated with major depression. Total score: 0 to 26; higher score indicates more depression.
Time Frame: Week 12
Population: Intent-to-treat (ITT) population included all enrolled participants. Here, 'N' (number of participants analyzed) signifies those participants who had data available and were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Hamilton Depression Scale (HAM-D): Participants who were administered Hamilton depression scales, HAM-D17 and HAM-D7.
Arm/Group | Hamilton Depression Scale (HAM-D)
Number analyzed (Participants) | 843
Percentage of participants | 54.4 [51.1 to 57.8]

2. Secondary Outcome: Percentage of Participants With Remission Based on Beck Depression Inventory (BDI)
Description: Remission according to BDI: BDI score less than (<) 10. BDI: 21 item participant rated inventory evaluates depression symptoms, cognition, and physical symptoms of fatigue, weight loss, lack of interest in sex. Individual items are scored on a 4 point scale (0 to 3), with 0=none/absent and 3=most severe. Total score: 0 to 63; higher score indicates more depression.
Time Frame: Week 12
Population: ITT population included all enrolled participants. Here, 'N' (number of participants analyzed) signifies those participants who had data available and were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Beck Depression Inventory (BDI): Participants who were administered BDI.
Arm/Group | Beck Depression Inventory (BDI)
Number analyzed (Participants) | 842
Percentage of participants | 64.6 [61.4 to 67.8]

3. Secondary Outcome: Hamilton Depression Scale 17 (HAM-D17), HAM-D7 and Beck Depression Inventory (BDI)
Description: HAM-D17: clinician-administered scale; assesses 17 items related to major depression (MD). Individual items scored on 3 point (0 to 2) or 5 point scale (0 to 4); 0=absent, 4=most severe. Total score: 0 to 66. HAM-D7: subset of HAM-D17; assesses 7 items related to MD. Total score: 0 to 26. BDI: 21 item participant rated inventory evaluates depression symptoms, cognition, physical symptoms of fatigue, weight loss, lack of interest in sex. Individual item scored on 4 point scale (0 to 3); 0=absent, 3=most severe. Total score: 0 to 63. For all the 3 scales, higher score represented more depression.
Time Frame: Baseline, Week 12
Population: ITT population included all enrolled participants. Here, 'N' (number of participants analyzed) signifies those participants who had data available at baseline and were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Hamilton Depression Scale (HAM-D17): Participants who were administered HAM-D17.
- Hamilton Depression Scale (HAM-D7): Participants who were administered HAM-D7, a subset of clinician-administered rating scale HAM-D17.
Arm/Group | Hamilton Depression Scale (HAM-D17) | Hamilton Depression Scale (HAM-D7) | Beck Depression Inventory (BDI)
Number analyzed (Participants) | 851 | 851 | 850
units on a scale
  Baseline | 25.18 (5.38) | 13.53 (3.22) | 31.45 (8.95)
  Week 12 | 7.31 (6.03) | 4.07 (3.51) | 9.03 (8.03)
  Change from baseline at Week 12 | 17.89 (6.74) | 9.48 (3.82) | 22.42 (10.02)
Statistical Analysis 1: Comparison: Hamilton Depression Scale (HAM-D17) vs Hamilton Depression Scale (HAM-D7); Change from baseline at Week 12: Pearson's correlation coefficient was used to evaluate compatibility between the questionnaires; Test type: Superiority or Other; p < 0.0001, Pearson's correlation — The statistical testing was done at alpha = 0.05; Pearson's correlation coefficient = 0.899, 95% CI 2-sided [0.886 to 0.911]
Statistical Analysis 2: Comparison: Hamilton Depression Scale (HAM-D17) vs Beck Depression Inventory (BDI); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Pearson's correlation — The statistical testing was done at alpha = 0.05; Pearson's correlation coefficient = 0.797, 95% CI 2-sided [0.771 to 0.820]
Statistical Analysis 3: Comparison: Hamilton Depression Scale (HAM-D7) vs Beck Depression Inventory (BDI); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Pearson's correlation — The statistical testing was done at alpha = 0.05; Pearson's correlation coefficient = 0.765, 95% CI 2-sided [0.736 to 0.791]

4. Secondary Outcome: Number of Participants With Residual Symptoms in Case of Non Remission
Description: Number of participants with residual symptoms who did not achieve remission was assessed. Remission according to HAM-D: HAM-D17 score =< 7 or HAM-D7 score =<3. Remission according to BDI: BDI score <10. HAM-D17: assessed 17 items associated with MD. Individual items scored on 3 point (0 to 2) or 5 point scale (0 to 4); 0=absent, 4=most severe. Total score: 0 to 66. HAM-D7: assessed 7 items associated with MD. Total score: 0 to 26. BDI assessed severity of depressive symptoms. Individual items are scored on a 4 point scale (0 to 3), with 0=none/absent and 3=most severe. The total score: 0 to 63. For all the 3 scales, higher score indicated more severe depression.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- All Participants: All participants diagnosed with major depressive disorder (MDD) who either started treatment with any anti-depressive agent for MDD for the first time or had a change in treatment as per physician's discretion and did not display remission.
Arm/Group | All Participants
Number analyzed (Participants) | 378
participants
  Emotional disorders | 59
  Sleep disorders | 35
  Behavioral disorders | 22
  Anxiety disorders | 22
  Psychosomatic disorders | 20
  Sexual disorders | 4
  No improvement | 3
  Psychotic disorders | 1

ADVERSE EVENTS:
Description: There were no adverse events collected in this observational non-interventional study.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Protocol did not indicate primary or secondary endpoints and designation of endpoints as primary or secondary endpoints was arbitrary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.